CLINICAL TRIAL: NCT06990555
Title: Cast Art for Kids With Extremity Fractures on Satisfaction and Perception of Pain (CAKEPOP)
Brief Title: Cast Art for Kids With Extremity Fractures
Acronym: CAKE POP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vanna Rocchi, PI, United States Naval Medical Center, Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 939056
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Fractures, Bone
Keywords: Cast; Art; Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — POLR1G protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neutral White Cast (Other): This intervention consists of receiving a cast of neutral white color.
  Interventions: Other: Neutral White Cast
- Color Wrapped Cast (Other): This intervention consists of receiving a cast of color that is the choice of the participant.
  Interventions: Other: Color Wrapped Cast
- Cast with Cast Art (Other): This intervention consists of receiving a cast with art at the request of the participant, to include drawing, multiple colors, glitter, and any artwork.
  Interventions: Other: Cast with Cast Art

INTERVENTIONS:
Other: Neutral White Cast — This intervention consists of receiving a cast of neutral white color.
  Arms: Neutral White Cast
Other: Color Wrapped Cast — This intervention consists of receiving a cast of color that is the choice of the participant.
  Arms: Color Wrapped Cast
Other: Cast with Cast Art — This intervention consists of receiving a cast with art at the request of the participant, to include drawing, multiple colors, glitter, and any artwork.
  Arms: Cast with Cast Art

SUMMARY:
The goal of this clinical trial is to compare casts with cast art versus those without art in children who sustain a fracture of the extremity. The main goals are:

* Determine the difference in satisfaction as measured by the visual analog scale for satisfaction between patients treated in a cast with cast customization versus those in a cast with no cast art
* Determine the difference in perceived pain scores between patients treated in a cast with cast customization versus those in a case with no cast art

Participants will be randomized to one of three groups: one with plain white cast, one with cast of color wrap of choice, and one with custom cast art.

Researchers will compare to see the differences in satisfaction and perception of pain based on what cast the study participant receives.

DETAILED DESCRIPTION:
Upper and lower extremity fractures are common amongst the pediatric population, with nearly 1 in every 5 children sustaining a fracture throughout their childhood and adolescence. Immobilization following an upper or lower extremity fracture is essential for treatment and bony healing, and this is most commonly performed with casting. Casts are placed in the acute setting in the emergency department or at an outpatient follow up visit; however, if the patient requires surgery, casts are also placed in the post operative period to aid in bony healing through immobilization. Length of treatment in the cast is dependent on the type of fracture the patient sustains, in addition to the bony healing that is analyzed via serial radiographs.

Given the prevalence of upper and lower extremity fractures among the pediatric population, overall patient and parent satisfaction is a key goal of treatment. While casting is extensively used at numerous pediatric orthopaedic centers, there is a paucity of information detailing patient reported outcome measures following casting. Typically casts are left to be either white in color or wrapped with a color of the patient's choice. Further customization of casts is now being popularized especially in social media, including drawing on the casts or applying decorative top-coat layers to the cast. However, there is little information detailing patient satisfaction and pain scores following casting with different techniques.

The purpose of this study is to: determine the difference in satisfaction as measured by the visual analog scale for satisfaction between patients treated in a cast with cast customization versus those in a cast with no cast art and (2) determine the difference in perceived pain scores between patients treated in a cast with cast customization versus those in a case with no cast art.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years old and greater, and less than 18 years old
* Sustained an upper or lower extremity fracture
* Scheduled for orthopedic clinic visit for injury evaluation
* Have radiographic and clinical data available for review

Exclusion Criteria:

* Age 18 years old or greater at the time of screening
* Patient/parents do not consent to being included in the study
* Underwent surgery

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for Satisfaction | 0-2 weeks post injury, 4-6 weeks, and 8-12 weeks (if indicated)
  VAS for satisfaction will be obtained of the patient and parent. The scale range is from no satisfaction (Lowest) to extreme satisfaction (highest). The parent and child place a mark on the line the best describes their satisfaction level.

SECONDARY OUTCOMES:
PedsQL Pediatric Pain Questionnaire | 0-2 weeks post injury, 4-6 weeks, and 8-12 weeks (if indicated)
  PedsQL Pediatric Pain Questionnaire will be obtained of the patient and parent. The scale range is from not hurting/no discomfort/no pain (least pain) to hurting a whole lot/very uncomfortable/severe pain (highest pain). The parent and child place a mark on the line the best describes their satisfaction level.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States